CLINICAL TRIAL: NCT03350685
Title: Detection and Characteristic of Whipple Diseases in the Great Britany
Acronym: WHO
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: WHO (29BRC17.0179)
Record Dates: First submitted 2017-11-17; First posted 2017-11-22 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Whipple Disease
MeSH Terms: conditions — Whipple Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Classic Whipple's disease (CWD): Classic Whipple's disease (CWD), defined as
  * duodenal biopsy positive by PAS/immunohistochemistry
  * or blood positive by PCR
- Focal Whipple's disease (FWD): Focal Whipple's disease (FWD), defined as
  * joint fluid positive by PCR
  * but duodenal biopsy negative by PAS/immunohistochemistry
- Chronic T. whipplei-associated arthritis (CTWA): Chronic T. whipplei-associated arthritis (CTWA) defined as chronic arthritis and
  * duodenal biopsy, stool, or saliva positive by PCR
  * duodenal biopsy negative by PAS/immunohistochemistry
  * joint fluid negative by PCR

SUMMARY:
Whipple's disease is a chronic systemic infection caused by ubiquitous bacterium Tropheryma wipplei on a genetic predisposition which should be considered in patients with recurrent episodes of seronegative arthritis, erosive or not, or inflammatory low back pain, chronic diarrhea, persistent fever, unexplained neurological signs, uveitis, endocarditis, and epithelioid granuloma.

Laboratory tests may show malabsorption, erythrocyte sedimentation rate and C-reactive protein elevation, anemia, thrombocytosis, eosinophilia and lymphopenia.

None of theses findings is specific and most patients have arthritis or low back pain mimicking rheumatoid arthritis and spondyloarthritis.

As the disease is rare, chance for positive polymerase chain reaction testing for Tropheryma whipplei is low in this context.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* patient with at least a screening test for Whipple'disease
* participation agreement,

Exclusion Criteria:

* No test for Whipple'disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis whipple's disease
Sampling Method: Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2018-02-09 (Actual)

PRIMARY OUTCOMES:
Number of patients diagnosed as whipple's disease | Day 0 ( Date of diagnostic)
  Diagnosis of Whipple's disease based on
  * at least one suggestive clinical finding
  * at least one test detecting T. Whipplei
  * diagnosis made by a specialist
  * a dramatic and persistent response to antibiotic therapy
    * Hydroxychloroquine 200mgx2 plus Doxycycline 100mgx2
    * or trimethoprim/sulfamethoxazole 800/160mg x2

SECONDARY OUTCOMES:
Number of test performed in each centre | Day 0 (Date of diagnostic)
  Number of diagnoses according to tests
  Patients will be divided into three groups
  Classic Whipple's disease (CWD), defined as :
  * duodenal biopsy positive by PAS/immunohistochemistry
  * or blood positive by PCR
  Focal Whipple's disease (FWD)
  * joint fluid positive by PCR
  * but duodenal biopsy negative by PAS/immunohistochemistry
  Chronic T. whipplei-associated arthritis (CTWA): chronic arthritis and
  * duodenal biopsy, stool, or saliva positive by PCR
  * duodenal biopsy negative by PAS/immunohistochemistry
  * joint fluid negative by PCR

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - CHU d'ANGERS, Angers
  - CHRU de Brest, Brest
  - CH le MAns, Le Mans
  - CHU de Nantes, Nantes
  - CH d'ORLEANS, Orléans
  - CHU de POITIERS, Poitiers
  - CHU de Rennes, Rennes
  - CHU de Tours, Tours